CLINICAL TRIAL: NCT04246151
Title: Oral Vancomycin Versus Probiotics Versus Placebo for Prevention of Clostridium Difficile Infection in Colonized Patients (Decency-RCT): A Randomized Controlled Pilot Trial
Brief Title: Oral Vancomycin Versus Probiotics Versus Placebo for Prevention of Clostridium Difficile Infection in Colonized Patients
Acronym: Decency-RCT
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No patients enrolled. Identification of patients in allocated timeframe was not feasible.
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DECENCY-RCT
Record Dates: First submitted 2020-01-20; First posted 2020-01-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-09

CONDITIONS: Clostridium Difficile Colonization; Clostridium Difficile Diarrhea
MeSH Terms: interventions — Vancomycin; Probiotics

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either a probiotic, oral vancomycin, or placebo in a parallel-group 1:1:1 design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding will be done in a double-blind fashion. The patients, their caregiver, and the investigator will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vancomycin & probiotic placebo (Experimental): Vancomycin 125 mg orally every 12 hours plus probiotic placebo orally every 12 hours for the duration of systematic antibiotic for a maximum of 21 days.
  Interventions: Drug: Vancomycin; Drug: Probiotic Placebo
- Probiotic & vancomycin placebo (Experimental): Culturelle probiotic 20 billion active units orally every 12 hours plus vancomycin placebo orally every 12 hours for the duration of systematic antibiotic for a maximum of 21 days.
  Interventions: Dietary Supplement: Culturelle; Drug: Vancomycin Placebo
- Probiotic placebo & vancomycin placebo (Placebo Comparator): Vancomycin placebo orally every 12 hours and Culturelle placebo orally every 12 hours for the duration of systematic antibiotic for a maximum of 21 days.
  Interventions: Drug: Vancomycin Placebo; Drug: Probiotic Placebo

INTERVENTIONS:
Drug: Vancomycin — Vancomycin capsules
  Other Names: JAMP-vancomycin
  Arms: Vancomycin & probiotic placebo
Dietary Supplement: Culturelle — Culturelle capsules
  Other Names: Lactobacillus rhamnosus GG
  Arms: Probiotic & vancomycin placebo
Drug: Vancomycin Placebo — sugar pill manufactured to mimic the vancomycin 125 mg capsule
  Other Names: Placebo for Vancomycin
  Arms: Probiotic & vancomycin placebo; Probiotic placebo & vancomycin placebo
Drug: Probiotic Placebo — sugar pill manufactured to mimic 10 billion unit probiotic capsules.
  Other Names: Placebo for probiotic
  Arms: Probiotic placebo & vancomycin placebo; Vancomycin & probiotic placebo

SUMMARY:
The goal of this pilot study is to assess the feasibility of randomizing hospitalized patients that are colonized with C. difficile and started on systemic antibiotics to either a probiotic, oral vancomycin, or placebo in a parallel-group 1:1:1 design. The ultimate goal is to conduct an appropriately-powered RCT to determine the optimal method for reducing C difficile infection in colonized patients.

DETAILED DESCRIPTION:
In this study, patients will be screened for C. difficile colonization

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18 years of age or older identified as asymptomatic carriers of C. difficile (i.e. not meeting case definition of C. difficile infection, see below)
* Started on systemic (oral or intravenous) antibiotics for any (presumed) bacterial infection
* Patient must have vitals (heart rate, blood pressure, temperature), estimated creatinine clearance (using the Chronic Kidney Disease Epidemiology equation (CKD-Epi)) and a complete blood count available within 24 hours of enrolment

Exclusion Criteria:

* On a course of systemic antibiotics that had been started more than 72 hours ago (as current evidence suggests that the earlier probiotics are started, the more efficacious they are)
* Patient with C. difficile, i.e. presence of diarrhea (three or more loose or watery stools within 24 hours), or fevers or hypotension from C. difficile infection
* Any patients with contra-indications to probiotics or vancomycin:

  * Immunosuppressed (primary or acquired immunodeficiency, including AIDS (defined as AIDS defining condition or cluster of differentiation 4 (CD4) nadir of <200/ul), hematologic malignancies, long-term systemic corticosteroid treatment, active treatment with chemotherapeutic agents or biologicals, autoimmune diseases, nephrotic syndrome)
  * Structural heart disease (e.g. atrial septal defect, ventricular septal defect)
  * Gastroesophageal or compromised gut integrity (e.g. short gut syndrome, intestinal injury or dysfunction, inflammatory bowel diseases including current or past history of Crohn's disease and ulcerative colitis)
  * Patients on systemic aminoglycosides, ethacrynic acid, polymixin B, or colistin.
  * Prior or current hearing loss
  * Female patients with known pregnancy or who are planning to get pregnant, or who are breastfeeding
  * Patients with end-stage renal diseases defined as an estimated glomerular filtration rate of <15ml/min, or absence of a current estimated creatinine clearance
  * History of an allergic reaction to one of the study drugs, or sensitivity to milk
* Patients started on probiotics or oral vancomycin while in hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Number of patients identified and randomized to a treatment arm within 72 hour of beginning a systematic antibiotic. | 1 year
  Feasibility will be assessed using the following parameters:
  Proportion of eligible participants screened that are randomized within 72 hours of antibiotic exposure (goal ≥ 90%)
  * Proportion of participants receiving all doses of study medication (goal ≥ 90%)
  * Proportion of participants with complete follow up at 14 days (goal ≥ 95%)
Development of C difficile associated diarrhea within 14 days of randomization | 1 year
  Development of C difficile associated diarrhea within 14 days of randomization to one of the treatment arms as defined by the Provincial Infectious Diseases Advisory Committee (PIDAC)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with researchers that are not directly involved in this study. Overall data will be shared in the context of peer reviewed journal publications or scientific presentations.